CLINICAL TRIAL: NCT04955808
Title: Early Onset Malignancies Initiative (EOMI): Molecular Profiling of Breast, Colon, Kidney, Liver, Multiple Myeloma, and Prostate Among Racially and Ethnically Diverse Populations
Brief Title: Biospecimen Collection in Identifying Genetic Changes in Patients With Breast, Prostate, Colorectal, Liver, or Kidney Cancer or Multiple Myeloma Undergoing Surgery
Status: Suspended | Type: Observational
Why Stopped: Due to slow accrual on this trial, we will allow sites time to work on close-out procedures and filling out necessary paperwork before taking the steps to forma
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NCI-2017-01572; NCI-2017-01572 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); DCP-002 (Other: National Cancer Institute Division of Cancer Prevention); DCP-002 (Other: DCP); DCP-002 (Other: CTEP)
Record Dates: First submitted 2021-07-08; First posted 2021-07-09 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Breast Carcinoma; Colon Carcinoma; Invasive Carcinoma; Kidney Carcinoma; Liver Carcinoma; Malignant Solid Neoplasm; Multiple Myeloma; Prostate Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Carcinoma, Renal Cell; Carcinoma, Hepatocellular; Multiple Myeloma; Prostatic Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue, blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ancillary-correlative (biospecimen collection): Patients undergo collection of tumor tissue during surgery. Patients also undergo blood samples. Samples collected may undergo genetic analysis including whole exome sequencing.
  Interventions: Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of tissue and blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This research trial studies how well biospecimen collection works in identifying genetic changes in patients with breast, prostate, colorectal, liver, or kidney cancer or multiple myeloma undergoing surgery. Studying samples collected during surgery may add to the understanding of cancer by looking for the genetic changes that cause early cancer onset in people of certain racial and ethnic groups.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To acquire tissue and blood, and other biospecimens for research purposes during procedures for clinical care to accelerate our understanding of the molecular basis of early onset cancers occurring in racial and/or ethnic minority populations through the application of genome analysis technologies, including large- scale genome sequencing and clinical data analysis.

OUTLINE:

Patients undergo collection of tumor tissue during surgery. Patients also undergo blood samples. Samples collected may undergo genetic analysis including whole exome sequencing.

After completion of study, patients are followed for up at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with either:

  * Histologically confirmed invasive carcinoma or multiple myeloma OR
  * Clinical diagnosis of carcinoma or multiple myeloma OR
  * Suspected clinical diagnosis of multiple myeloma
* Patients with one of following tumor types and age ranges:

  * Breast cancer diagnosis at ages 18-45
  * Colon cancer diagnosis at ages 18-55
  * Kidney cancer at diagnosis at ages 18-50 (American Indian or Alaska Native [AIAN] and non-Hispanic Whites [NHW] only)
  * Liver cancer diagnosis at ages 18-55
  * Prostate cancer diagnosis at ages 18-55
  * Multiple myeloma diagnosis at ages 18-50
* Patients whose tumor specimen was collected or will be collected during one of the following routine procedures:

  * Surgery to remove cancer OR
  * Routine biopsy procedures performed to confirm a histologic diagnosis OR
  * Routine biopsy procedure performed to obtain additional tumor material for routine prognostic or predictive biomarkers OR
  * Routine procedure to place a vascular access device prior for systemic therapy
* Patients who have received no therapy for their cancer other than surgery, irrespective of stage
* Collection of specimens from living patients:

  * Ability to understand and willingness to sign a written informed consent document indicating their willingness to have their tissue or biologic fluid specimens used for research as outlined in this protocol
* Collection of specimens from deceased patients:

  * Banked tissue samples and/or banked biologic fluid specimens of deceased patients may be used as long as all samples or specimens are properly de- identified prior to submission
* Sites must use the Central Institutional Review Board for the National Cancer Institute (NCI CIRB).

Exclusion Criteria:

* Patients who do not meet criteria for an early onset malignancy
* Prior systemic therapy or radiation therapy for their malignancy
* Tumor does not meet quality metrics
* Patient refused consent for use of tissue for research activities included in the Early Onset Malignancies Initiative
* A diagnosis of a synchronous invasive malignancy
* Patients with a history of invasive cancer or hematologic malignancy in preceding 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery to remove tumor tissue
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2017-02-07 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Acquisition of tissue, blood, and other biospecimens for research purposes | Up to 3 years
  Will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Bennett, Principal Investigator — National Cancer Institute Division of Cancer Prevention
Locations (1):
- National Cancer Institute Division of Cancer Prevention, Rockville, Maryland, United States